CLINICAL TRIAL: NCT02740972
Title: A Phase II, Dose Finding Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of NS-065/NCNP-01 in Boys With Duchenne Muscular Dystrophy (DMD)
Brief Title: Safety and Dose Finding Study of NS-065/NCNP-01 in Boys With Duchenne Muscular Dystrophy (DMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NS Pharma, Inc. (Industry)
Collaborators: Nippon Shinyaku Co., Ltd. (Industry); Cooperative International Neuromuscular Research Group (Network); Therapeutic Research in Neuromuscular Disorders Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NS-065/NCNP-01-201
Record Dates: First submitted 2016-03-23; First posted 2016-04-15 (Estimated); Results first posted 2021-07-12 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NS-065/NCNP-01 40mg/kg (Experimental): Six patients with confirmed DMD with genetic deletions amenable to exon 53 skipping will be administered an intravenous infusion of NS-065/NCNP-01 40mg/kg dose once a week for 24 weeks
  Interventions: Drug: NS-065/NCNP-01
- NS-065/NCNP-01 80mg/kg (Experimental): Six patients with confirmed DMD with genetic deletions amenable to exon 53 skipping will be administered an intravenous infusion of NS-065/NCNP-01 80mg/kg once a week for 24 weeks
  Interventions: Drug: NS-065/NCNP-01
- Placebo (Placebo Comparator): Two patients in each of the dose groups will be administered placebo as an intravenous infusion once a week for 4 weeks followed by 20 weeks of open label treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NS-065/NCNP-01
  Arms: NS-065/NCNP-01 40mg/kg; NS-065/NCNP-01 80mg/kg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The main objective of this study is to evaluate the safety of a high (80mg/kg) and low (40mg/kg) dose of NS-065/NCNP-01 delivered as an intravenous infusion in patients with Duchenne Muscular Dystrophy (DMD) amendable to exon 53 skipping. Additional objectives include tolerability, muscle function and strength, pharmacokinetics and pharmacodynamics.

DETAILED DESCRIPTION:
This is a Phase II, multiple center, 2-period, randomized, placebo-controlled, dose finding study of NS-065/NCNP-01 administered by infusion once weekly for 24 weeks to ambulant boys ages 4-<10 years with DMD. Two dose level cohorts will be enrolled. Period 1 of this study will be conducted in a double-blind fashion. Randomized patients will receive weekly IV infusions of NS-065/NCNP-01 or placebo for the first 4 weeks of their participation (Period 1) and NS-065/NCNP-01 by IV infusion for weeks 5-24 (20 weeks of active treatment - Period 2). Analysis of safety data from Period 1 of the 40mg/kg dose cohort will be completed prior to enrolling patients in the 80mg/kg dose cohort.

Patients completing the 24-week study will be eligible for an open-label extension study.

Clinical efficacy will be assessed at regularly scheduled study visits, including functional tests such as the six-minute walk test (6MWT), time to stand (TTSTAND), time to run/walk 10 meters (TTRW), time to climb 4 stairs (TTCLIMB) and quantitative muscle testing (QMT). All patients will undergo a muscle biopsy of the bicep at baseline and a second muscle biopsy at Week 24.

Safety will be assessed through the collection of adverse events (AEs), blood and urine laboratory tests, electrocardiograms (ECGs), vital signs, and physical examinations throughout the study.

Serial blood samples will be taken at four of the study visits to assess the pharmacokinetics of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥ 4 years and <10 years of age
* Confirmed DMD mutation(s) in the dystrophin gene that is amenable to skipping of exon 53 to restore the dystrophin mRNA reading frame;
* Able to walk independently without assistive devices;
* Ability to complete the time to stand, time to run/walk and time to climb assessments;
* Stable dose of glucocorticoid for at least 3 months

Exclusion Criteria:

* Acute illness within 4 weeks prior to the first dose of study medication;
* Evidence of symptomatic cardiomyopathy. [Note: Asymptomatic cardiac abnormality on investigation would not be exclusionary];
* Severe allergy or hypersensitivity to medications;
* Severe behavioral or cognitive problems that preclude participation in the study, in the opinion of the Investigator;
* Previous or ongoing medical condition, medical history, physical findings or laboratory abnormalities that could affect safety, make it unlikely that treatment and follow-up will be correctly completed or impair the assessment of study results, in the opinion of the Investigator;
* Patient is taking any other investigational drug currently or within 3 months prior to the start of study treatment; or
* Patient has had surgery within the 3 months prior to the first anticipated administration of study medication or surgery is planned for anytime during the duration of the study;
* Patient has previously participated in this study or any other study during which NS-065/NCNP-01 was administered.

Ages: 4 Years to 9 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula R. Clemens, MD, Study Chair — University of Pittsburgh
Locations (7):
- United States (6):
  - UC Davis, Sacramento, California
  - University of Florida Health, Gainesville, Florida
  - Lurie Children's Hospital, Chicago, Illinois
  - Washington University, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Richmond at VCU, Richmond, Virginia
- Alberta Children's Hospital, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Clemens PR, Rao VK, Connolly AM, Harper AD, Mah JK, Smith EC, McDonald CM, Zaidman CM, Morgenroth LP, Osaki H, Satou Y, Yamashita T, Hoffman EP; CINRG DNHS Investigators. Safety, Tolerability, and Efficacy of Viltolarsen in Boys With Duchenne Muscular Dystrophy Amenable to Exon 53 Skipping: A Phase 2 Randomized Clinical Trial. JAMA Neurol. 2020 Aug 1;77(8):982-991. doi: 10.1001/jamaneurol.2020.1264. PMID 32453377

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment occurred between December 16, 2016, and August 17, 2017, at 6 sites in the US and Canada.
Pre-assignment Details: A total of 17 patients were screened at 6 sites in the United States and Canada. Of the 17 patients screened, 1 failed to meet an inclusion criterion.
Groups:
- Placebo (Period 1); NS-065/NCNP-01 40mg/kg (Period 1); NS-065/NCNP-01 80mg/kg (Period 1): 4-week Double-blinded placebo-controlled period (Period 1) Week 0 - Week 4
- NS-065/NCNP-01 40mg/kg (Period 2); NS-065/NCNP-01 80mg/kg (Period 2): 20-week Open-label treatment period (Period 2) Week 5 - Week 24
Period: 4-week Double-blinded Placebo-controlled
Arm/Group | Placebo (Period 1) | NS-065/NCNP-01 40mg/kg (Period 1) | NS-065/NCNP-01 80mg/kg (Period 1) | NS-065/NCNP-01 40mg/kg (Period 2) | NS-065/NCNP-01 80mg/kg (Period 2)
Started | 5 | 6 | 5 | 0 | 0
Completed | 5 | 6 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: 20-week Open Label Treatment Period
Arm/Group | Placebo (Period 1) | NS-065/NCNP-01 40mg/kg (Period 1) | NS-065/NCNP-01 80mg/kg (Period 1) | NS-065/NCNP-01 40mg/kg (Period 2) | NS-065/NCNP-01 80mg/kg (Period 2)
Started | 0 | 0 | 0 | 8 | 8
Completed | 0 | 0 | 0 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 16 participants were enrolled and 8 participants participated in each of the 2 dose cohorts.
Groups:
- NS-065/NCNP-01 40mg/kg: Patients with confirmed DMD with genetic deletions amenable to exon 53 skipping will be administered an intravenous infusion of NS-065/NCNP-01 40mg/kg once a week for 24 weeks
- NS-065/NCNP-01 80mg/kg: Patients with confirmed DMD with genetic deletions amenable to exon 53 skipping will be administered an intravenous infusion of NS-065/NCNP-01 80mg/kg once a week for 24 weeks
- Total: Total of all reporting groups
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.5 (1.8) | 7.2 (2.0) | 7.4 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 6 | 14
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 23.7 (4.7) | 22.3 (6.2) | 23.0 (5.3)
Height [Mean (Standard Deviation); unit: cm] | 114.6 (6.5) | 112.2 (10.0) | 113.4 (8.2)
Body Mass Index(BMI) [Mean (Standard Deviation); unit: kg/m^2] | 17.9 (2.3) | 17.4 (2.0) | 17.7 (2.1)
Time to run/walk 10m velocity [Mean (Standard Deviation); unit: m/s] | 1.67 (0.39) | 1.88 (0.36) | 1.77 (0.37)
Time to run/walk 10m [Mean (Standard Deviation); unit: second] | 6.30 (1.59) | 5.55 (1.34) | 5.93 (1.47)
Time to stand from supine velocity [Mean (Standard Deviation); unit: rise/s] | 0.26 (0.06) | 0.25 (0.09) | 0.25 (0.07)
Time to stand from supine [Mean (Standard Deviation); unit: second] | 4.17 (1.15) | 4.76 (2.58) | 4.44 (1.96)
6-Minute walk test [Mean (Standard Deviation); unit: m] | 391.4 (33.3) | 353.4 (106.3) | 372.4 (78.6)
Time to climb 4 stairs velocity [Mean (Standard Deviation); unit: m/s] | 0.27 (0.08) | 0.32 (0.08) | 0.30 (0.08)
Time to climb 4 stairs [Mean (Standard Deviation); unit: second] | 3.90 (0.93) | 3.33 (0.94) | 3.61 (0.95)
NSAA score [Mean (Standard Deviation); unit: scores on a scale] — The NSAA is a functional scale devised for use in ambulant children with Duchenne muscular dystrophy (DMD). It consists of 17 activities graded 0 (unable to perform), 1 (performs with modifications), 2 (normal movement). It assesses abilities necessary to remain ambulant that have been found to progressively deteriorate in untreated DMD patients, as well as in other muscular dystrophies such as Becker Muscular Dystrophy. NSAA Total Score ranges from 0 to 34, with a score of 34 implying normal function.
  scores on a scale | 24.8 (5.9) | 23.8 (5.1) | 24.3 (5.4)
Dystrophin Production by Western Blot [Mean (Standard Deviation); unit: % of normal control levels]
  Normalized to Myosin | 0.3 (0.10) | 0.6 (0.82) | 0.4 (0.60)
  Normalized to Alpha-Actinin | 0.2 (0.22) | 0.4 (0.67) | 0.3 (0.50)
Dystrophin Production by Mass Spectrometry [Mean (Standard Deviation); unit: % of normal control levels] | 0.5 (0.15) | 0.6 (0.19) | 0.6 (0.17)
Dystrophin Production by Immunofluorescence [Mean (Standard Deviation); unit: % of normal control levels] | 1.5 (0.98) | 1.8 (2.36) | 1.7 (1.75)
Dystrophin Production by RT-PCR for mRNA - Percentage of Exons Skipped - Molarity [Mean (Standard Deviation); unit: % of normal control levels] | 0.0 (0.00) | 0.0 (0.00) | 0.0 (0.00)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events as Assessed by CTCAE v4.0.
Description: Treatment emergent adverse events (TEAEs) were summarized for Period 1 by comparing low dose to high dose to placebo and for Period 2 between the low dose cohort and the high dose cohort. TEAEs were summarized both at the patient level for number of TEAEs, highest severity, relationship, action and outcome and at the TEAE level (summarizing events) by organ system and preferred term TEAE as well as severity, relationship, action and outcome.
  The Medical Dictionary for Regulatory Activities (MedDRA) version 20.1 was used and the Common Terminology Criteria for Adverse Events (CTCAE) grading.
Time Frame: 24 weeks of treatment
Population: Within each category, patients were counted only once if they had >1 event reported during the treatment period.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (Period 1): 4-week Double-blinded placebo-controlled period (Period 1)
  Two patients in each of the dose groups will be administered placebo as an intravenous infusion once a week for 4 weeks followed by 20 weeks of open label treatment
- NS-065/NCNP-01 40mg/kg (Period 1); NS-065/NCNP-01 80mg/kg (Period 1): 4-week Double-blinded placebo-controlled period (Period 1)
- NS-065/NCNP-01 40mg/kg (Period 2); NS-065/NCNP-01 80mg/kg (Period 2): 20-week Open-label treatment period (Period 2)
Arm/Group | Placebo (Period 1) | NS-065/NCNP-01 40mg/kg (Period 1) | NS-065/NCNP-01 80mg/kg (Period 1) | NS-065/NCNP-01 40mg/kg (Period 2) | NS-065/NCNP-01 80mg/kg (Period 2) | Total
Number analyzed (Participants) | 5 | 6 | 5 | 8 | 8 | 16
Participants
  Participants with TEAE | 3 | 4 | 4 | 5 | 7 | 15
  Participants with drug-related TEAE | 0 | 0 | 0 | 0 | 0 | 0
  Participants with CTCAE ≥ Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  Participants with TEAEs leading to discontinuation | 0 | 0 | 0 | 0 | 0 | 0
  Participants with serious TEAE | 0 | 0 | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Dystrophin Production by Western Blot
Description: Percentage normal dystrophin production in muscle biopsies from study participants at baseline and after 24 weeks treatment was measured by Western blot.
  To analyze dystrophin induction, biopsies were taken from a biceps muscle at baseline and the other biceps muscle after 24 weeks of treatment. Muscle samples were snap frozen and delivered to a central laboratory. All laboratory researchers remained blinded to sample identity. Dystrophin protein levels were assessed using standard curves on each gel (range from 0-25% of normal levels) generated by mixing 5 normal control samples with one DMD sample.
Time Frame: Baseline and 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: % of normal control levels
Groups:
- NS-065/NCNP-01 40mg/kg: NS-065/NCNP-01 40mg/kg dose once a week for 20-24 weeks
- NS-065/NCNP-01 80mg/kg: NS-065/NCNP-01 80mg/kg dose once a week for 20-24 weeks
- Total NS-065/NCNP-01 Group: Of the 16 patients randomized, all patients received treatment with NS-065/NCNP-01 and all patients completed treatment with NS-065/NCNP-01.
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
% of normal control levels
  Normalized to Myosin | 5.7 (2.37) | 5.9 (4.50) | 5.8 (3.47)
  Normalized to Alpha-Actinin | 5.4 (2.79) | 3.7 (2.37) | 4.5 (2.64)

3. Secondary Outcome: Dystrophin Production by RT-PCR for mRNA - Percentage of Exons Skipped - Molarity
Description: The alteration of mRNA splicing was measured by RT-PCR of dystrophin mRNA transcripts from a patient muscle biopsy at baseline and after 24 weeks treatment.
  To analyze dystrophin induction, biopsies were taken from a biceps muscle at baseline and the other biceps muscle after 24 weeks of treatment. Muscle samples were snap frozen and delivered to a central laboratory. All laboratory researchers remained blinded to sample identity. For RT-PCR, bands corresponding to specific versions of the spliced dystrophin mRNA were visualized by gel electrophoresis, and the amounts of different mRNA isoforms were compared.
Time Frame: Baseline and 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: % of normal control levels
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
% of normal control levels | 17.4 (7.17) | 43.9 (16.68) | 30.6 (18.45)

4. Secondary Outcome: Dystrophin Production by Mass Spectrometry
Description: The production of dystrophin protein was measured by stable isotope mass spectrometry methods from a patient muscle biopsy at baseline and after 24 weeks treatment.
  To analyze dystrophin induction, biopsies were taken from a biceps muscle at baseline and the other biceps muscle after 24 weeks of treatment. Muscle samples were snap frozen and delivered to a central laboratory. All laboratory researchers remained blinded to sample identity.
  Dystrophin peptides were identified and quantified using reversed-phase nanoflow high-performance liquid chromatography with high resolution Mass Spectrometry.
Time Frame: Baseline and 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: % of normal control levels
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
% of normal control levels | 2.1 (1.09) | 4.2 (3.73) | 3.1 (2.88)

5. Secondary Outcome: Dystrophin Production by Immunofluorescence
Description: The production of dystrophin protein was measured by immunofluorescence staining methods from a patient muscle biopsy at baseline and after 24 weeks treatment.
  To analyze dystrophin induction, biopsies were taken from a biceps muscle at baseline and the other biceps muscle after 24 weeks of treatment. Muscle samples were snap frozen and delivered to a central laboratory. All laboratory researchers remained blinded to sample identity.
  Immunofluorescence staining for dystrophin was performed on serial muscle biopsy sections in duplicate.
Time Frame: Baseline and 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: % dystrophin-positive fibers
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
% dystrophin-positive fibers | 14.2 (7.77) | 34.8 (20.42) | 24.5 (18.32)

6. Secondary Outcome: Change From Baseline in Muscle Strength as Measured by Quantitative Muscle Testing (QMT).
Description: A secondary efficacy endpoint was compared to Pre-Infusion Visit: quantitative muscle testing (QMT).
Time Frame: Baseline and 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: lb
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
lb
  Handgrip | -0.2029 (2.98334) | -0.8513 (1.85797) | -0.4808 (2.49621)
  Dominant Side Handgrip | -0.4173 (2.46596) | -1.0867 (1.75915) | -0.7041 (2.14074)
  Non-Dominant Side Handgrip | -0.2280 (3.39211) | -0.1780 (2.27428) | -0.2066 (2.86108)
  Elbow Flexors (biceps) | 0.3190 (1.99880) | -0.7110 (1.61528) | -0.1224 (1.85326)
  Dominant Side Elbow Flexors (biceps) | 0.5111 (2.57829) | -0.4468 (1.49138) | 0.1006 (2.16263)
  Non-Dominant Side Elbow Flexors (biceps) | 0.2067 (2.71502) | -0.3732 (2.50228) | -0.0163 (2.54427)
  Elbow Extensors (triceps) | 0.6777 (2.65006) | 0.6895 (1.00990) | 0.6828 (2.04299)
  Dominant Side Elbow Extensors (triceps) | 0.7046 (2.78271) | 0.6502 (0.81291) | 0.6813 (2.10345)
  Non-Dominant Side Elbow Extensors (triceps) | 0.0001 (2.34657) | 0.5168 (1.44498) | 0.2216 (1.95920)
  Knee Flexors (hamstrings) | -1.2209 (3.37401) | -0.0283 (3.43240) | -0.7098 (3.32207)
  Dominant Side Knee Flexors (hamstrings) | -1.8985 (4.01798) | -0.7175 (3.64572) | -1.3924 (3.76469)
  Non-Dominant Side Knee Flexors (hamstrings) | -1.7373 (3.10626) | 0.6377 (2.03566) | -0.7194 (2.87696)
  Knee Extensors (quadriceps) | -2.2261 (4.82146) | 1.5798 (3.33316) | -0.5950 (4.53990)
  Dominant Side Knee Extensors (quadriceps) | -2.1524 (4.58595) | 2.0867 (2.96796) | -0.3356 (4.41039)
  Non-Dominant Side Knee Extensors (quadriceps) | -0.5994 (4.38150) | 1.3308 (4.44474) | 0.2279 (4.34950)

7. Secondary Outcome: Change From Baseline in Distance Traveled in the Six-Minute Walk Test (6MWT).
Description: A secondary efficacy endpoint was compared to Pre-Infusion Visit: Six-Minute Walk Test (6MWT).
Time Frame: Baseline and 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: m
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
m | 15.6 (26.40) | 44.0 (41.98) | 28.9 (36.31)

8. Secondary Outcome: Change From Baseline in Time to Climb 4 Stairs (TTCLIMB).
Description: A secondary efficacy endpoint was compared to Pre-Infusion Visit: Time to Climb 4 Stairs (TTCLIMB).
Time Frame: Baseline and 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: second
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
second | -0.34 (1.140) | 0.00 (0.600) | -0.17 (0.897)

9. Secondary Outcome: Change From Baseline in Time to Climb 4 Stairs (TTCLIMB) Velocity
Description: A secondary efficacy endpoint was compared to Pre-Infusion Visit: Time to Run/Walk 10 meters (TTRW). The results were converted into velocity (meter/time).
Time Frame: Baseline and 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
m/s | 0.07 (0.105) | -0.00 (0.054) | 0.32 (0.088)

10. Secondary Outcome: Change From Baseline in Time to Run/Walk 10 Meters (TTRW).
Description: A secondary efficacy endpoint was compared to Pre-Infusion Visit: Time to Run/Walk 10 meters (TTRW).
Time Frame: Baseline and 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: second
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
second | -0.65 (1.225) | -0.66 (0.921) | -0.66 (1.047)

11. Secondary Outcome: Change From Baseline in Time to Run/Walk 10 Meters (TTRW) Velocity.
Description: as for outcome 9
Time Frame: Baseline and 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
m/s | 0.21 (0.291) | 0.24 (0.222) | 0.23 (0.251)

12. Secondary Outcome: Change From Baseline in Time to Stand (TTSTAND)
Description: A secondary efficacy endpoint was compared to Pre-Infusion Visit: Time to Stand (TTSTAND)
Time Frame: Baseline and 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: second
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
second | 0.05 (1.446) | -0.44 (0.750) | -0.19 (1.141)

13. Secondary Outcome: Change From Baseline in Time to Stand (TTSTAND) Velocity
Description: A secondary efficacy endpoint was compared to Pre-Infusion Visit: Time to Stand (TTSTAND).The results were converted into velocity (rise/time).
Time Frame: Baseline and 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: rise/time
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
rise/time | 0.02 (0.093) | 0.02 (0.060) | 0.02 (0.075)

14. Secondary Outcome: Change From Baseline in North Star Ambulatory Assessment (NSAA) Score.
Description: The NSAA is a functional scale devised for use in ambulant children with Duchenne muscular dystrophy (DMD). It consists of 17 activities graded 0 (unable to perform), 1 (performs with modifications), 2 (normal movement). It assesses abilities necessary to remain ambulant that have been found to progressively deteriorate in untreated DMD patients, as well as in other muscular dystrophies such as Becker Muscular Dystrophy. NSAA Total Score ranges from 0 to 34, with a score of 34 implying normal function.
Time Frame: Baseline and 24 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NS-065/NCNP-01 40mg/kg | NS-065/NCNP-01 80mg/kg | Total NS-065/NCNP-01 Group
Number analyzed (Participants) | 8 | 8 | 16
score on a scale | 0.5 (3.07) | 1.1 (2.80) | 0.8 (2.86)

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Incidence of Adverse Events as assessed by CTCAE v4.0
Groups:
- Placebo (Period 1): 4-week Double-blinded placebo-controlled period (Period 1) Week 0 - Week 4
  Two patients in each of the dose groups will be administered placebo as an intravenous infusion once a week for 4 weeks followed by 20 weeks of open label treatment
Arm/Group | Placebo (Period 1) | NS-065/NCNP-01 40mg/kg (Period 1) | NS-065/NCNP-01 80mg/kg (Period 1) | NS-065/NCNP-01 40mg/kg (Period 2) | NS-065/NCNP-01 80mg/kg (Period 2) | Total
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/5 | 0/8 | 0/8 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/5 | 0/8 | 0/8 | 0/16
Other Adverse Events (participants affected / at risk) | 3/5 | 4/6 | 4/5 | 5/8 | 7/8 | 15/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Period 1) (N=5) | NS-065/NCNP-01 40mg/kg (Period 1) (N=6) | NS-065/NCNP-01 80mg/kg (Period 1) (N=5) | NS-065/NCNP-01 40mg/kg (Period 2) (N=8) | NS-065/NCNP-01 80mg/kg (Period 2) (N=8) | Total (N=16)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 2 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 2
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Molluscum contagiosum (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 4 | 4
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Infusion site discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Injection site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Thirst (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 2
Abnormal behaviour (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The most restrictive relevant agreement on the PI provides that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is not less than 30 days from the time submitted to the sponsor for review.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/72/NCT02740972/Prot_SAP_000.pdf